CLINICAL TRIAL: NCT06725979
Title: Effect of the Rapid Palatal Expansion Treatment on Reported Sleeping Disorders in Children
Brief Title: Effect of the Palatal Expansion Treatment on Reported Sleeping Disorders in Children
Acronym: RPE PSQ HR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rijeka (Other)
Collaborators: University of Rijeka Faculty of Dental Medicine (Unknown)
Responsible Party: Principal Investigator, Visnja Katic, Assistant Professor, University of Rijeka
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: RPE PSQ; uniri-iskusni-biomed-23-36 (Other Grant/Funding Number: University of Rijeka)
Record Dates: First submitted 2024-12-05; First posted 2024-12-10 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-07

CONDITIONS: Narrow Maxilla
Keywords: palatal expansion; PSQ; facial scan; orthodontics; hyrax expander

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rapid maxillary expansion group (Active Comparator): expansion of the maxilla with hyrax expander
  Interventions: Device: maxillary expansion using hyrax expander
- control (No Intervention): no need for the maxillary expansion

INTERVENTIONS:
Device: maxillary expansion using hyrax expander — The rapid expansion of the upper jaw will be performed using palatal expander with hyrax screw, which will be activated 2x a day, until the needed width is reached (according to the cast analysis).
  Other Names: rapid palatal expansion
  Arms: Rapid maxillary expansion group

SUMMARY:
The goal of this clinical trial is to see if expanding the upper jaw with orthodontic therapy can help improve sleep related breathing problems in children. Parents or caregivers will complete the Pediatric Sleep Questionnaire (PSQ) to assess their child's sleep before and after treatment.

The study will include 20 children with a narrow upper jaw, and a control group of children without this condition. The main questions it aims to answer are:

* Will the 3D scans show significant changes in the face after therapy?
* Will the dental scans show a larger palate volume after treatment?
* Will parents/caregivers notice an improvement in their children's sleep problems after therapy? Researchers will compare 3D facial and dental scans, as well as PSQ results, before and one year after therapy to see if the treatment makes a difference.

Participants will:

* Receive orthodontic treatment to expand the upper jaw.
* Have their sleep related breathing problems assessed by parents or caregivers using the PSQ before and after treatment.
* Have 3D scans of their face and teeth taken before and after treatment.

DETAILED DESCRIPTION:
This comprehensive clinical study focuses on evaluating the therapeutic impact of orthodontic maxillary expansion treatment on sleep disorder assessments in children, as reported by their parents or guardians using the Pediatric Sleep Questionnaire (PSQ). Maxillary transverse constriction is a developmental disorder that can adversely affect the orofacial region, potentially influencing breathing patterns during sleep. The primary objective is to investigate whether orthodontic intervention to widen the upper jaw can lead to favorable developmental outcomes in the orofacial region and potentially alleviate sleep-related breathing disorders.

The study will involve 20 patients diagnosed with transverse maxillary constriction, identified through 3D scans of their face and dentition, compared against a control group of individuals without such constriction. Before and one year after treatment, participants will undergo 3D scanning of their facial structure and dentition, complemented by the completion of PSQ questionnaires by their parents or guardians. The study's hypotheses propose that following treatment, there will be notable changes in the mid-facial region evident from 3D facial scans, an increase in palate volume as indicated by dental scans, and a moderate improvement in reported sleep disorder symptoms based on parental observations.

The research methodology incorporates non-invasive 3D facial scanning technology, a methodological advancement that allows for precise assessment of facial changes pre-treatment and post-treatment. This approach contrasts with traditional 2D imaging, offering more detailed and accurate data on structural alterations. The study also highlights the utility of PSQ as a validated tool for evaluating sleep disorders in children, avoiding the need for expensive polysomnography.

By utilizing advanced imaging techniques and validated questionnaires, researchers seek to objectively measure treatment outcomes and correlate them with improvements in sleep quality and respiratory function. The study will utilize specialized equipment such as the Bellus 3D facial scanner and the Audaxceph software.

Ultimately, this study aims to enhance our understanding of the relationship between maxillary expansion therapy and sleep disorder improvement in children, potentially paving the way for optimized treatment protocols and improved patient outcomes sleep related breathing problems.

ELIGIBILITY:
Inclusion Criteria:

narrow maxilla

Exclusion Criteria:

hypodontia, craniodentofacial deformity-

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-04-08 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Facial scan | from enrollment to the end of treatment at one year on average
  3D facial scan of the surface of the face using stereo-photography
Dental scan | from enrollment to the end of treatment at one year on average
  3D scan of dentition
PSQ questionnaire | from enrollment to the end of treatment at one year on average
  Pediatric Sleep Questionnaire (PSQ) filled by the parents / caregivers

SECONDARY OUTCOMES:
Latero-lateral cephalogram | from enrollment to the end of treatment at one year on average
  Cranio-dento-facial characteristics as measured on latero-lateral cephalogram

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dental Medicine, Rijeka, Primorje-Gorski Kotar County, Croatia

IPD SHARING:
Plan to Share IPD: Undecided
IPD contains identifiable biometric data, and will be disclosed only on reasonable request.